CLINICAL TRIAL: NCT04058743
Title: Effect of Nickel Sensitivity on Patient Reported Outcomes After Total Knee Arthroplasty
Brief Title: Nickel Sensitivity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have decided to stop the study due to lack of enrollment
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, Professor of Orthopaedic Surgery, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18112703
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Knee Arthropathy; Allergic Reaction
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial with two groups: Total knee replacement with standard cobalt chromium components vs Total Knee Replacements with nickel free components.
Who Masked: Participant
Masking Description: Patients will be blinded to the type of implant that they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TKA with standard cobalt chromium components (Active Comparator): Patients randomized to this group will receive the standard cobalt chromium components in their total knee arthroplasty
  Interventions: Device: TKA with standard cobalt chromium components
- TKA with nickel free components (Experimental): Patients randomized to this group will receive nickel free components in their total knee arthroplasty
  Interventions: Device: TKA with nickel free components

INTERVENTIONS:
Device: TKA with nickel free components — Patients will be randomized to receive either the standard cobalt chromium components or nickel free components
  Arms: TKA with nickel free components
Device: TKA with standard cobalt chromium components — Patients will be randomized to receive either the standard cobalt chromium components or nickel free components
  Arms: TKA with standard cobalt chromium components

SUMMARY:
The purpose of this study is to compare clinical outcomes of patients with self reported nickel sensitivity undergoing primary total knee arthroplasty (TKA) with conventional, standard-of-care vs nickel-free implants. The hypothesis is that patients with a self-reported nickel sensitivity will have similar patient reported outcome scores compared to those patients without reported nickel sensitivity. Therefor the anticipation is for there to be no differences in other clinical outcome measures or functional outcome scores between the two cohorts.

DETAILED DESCRIPTION:
Metal implants are a mainstay of orthopedic treatment, and a variety of metal implants have been utilized for more than 40 years. Total knee replacement implants have been comprised of a variety of metal, ceramic, and plastic components. Current standard-of-care for TKA employs a cobalt chrome alloy femoral implant that articulates with the polyethylene surface of the tibial component. This cobalt chrome alloy can contain up to 1% nickel.

While most patients report pain relief and satisfaction after TKA, there are a number of complications that can result. Infection, component loosening, polyethylene wear, and malalignment are common reasons for persistent pain after TKA. Metal sensitivity as a cause of persistent pain after total joint arthroplasty is a controversial topic. Cutaneous metal hypersensitivity has a prevalence of approximately 10-15% in the general population, with nickel being the most common metal sensitizer with a prevalence near 14%. Cross reactivity with cobalt chrome and nickel is very common.

The role of metal allergy in orthopedic surgery and total joint arthroplasty is a poorly understood relationship. The cause and effect relationship of this process has not been delineated - it is unclear if the immunogenic response causes implant failure, or implant failure releases hapten particles with lead to a deep tissue reaction.

Metal hypersensitivity after TKA is a rarely documented phenomenon without specific diagnostic criteria, and there is much debate on if this is even a true diagnosis. The two most commonly described presentations include 1) dermatitis or 2) persistent painful synovitis although these have only been described in case reports without defined diagnostic criteria. Few reports exist regarding the diagnosis and management of these conditions. There is no reliable or generally accepted test to predict allergy to total joint replacement components. Patient history of metal sensitivity is not a reliable indicator of TJA outcome, as 25% of patients with well-functioning TJA implants have a reported metal allergy. A nickel or metal sensitivity has not been statistically identified as a risk factor for any specific cutaneous or deep tissue reaction, complication, or poor outcome after TKA.

Typically, metal sensitivity patients are identified after having a superficial skin reaction after dermal contact with a metal. Nickel containing jewelry is a common precipitator. The true diagnosis of skin sensitivity to metal is diagnosed by cutaneous patch testing, often employed by dermatologists. This test is not specific or sensitive for the diagnosis of deep tissue metal sensitivity. In a case control study, Granchi et al followed 94 patients without metal implants, with stable painless TKA, and with TKA and evidence of loosening. The study found no predictive value in dermal patch testing for metal hypersensitivity and the stability of TKA implants. Verma et al followed 30 patients with dermatitis following TKA. Fifteen were available for patch testing, but only seven patients tested 1+ or 2+ reaction to a metal. Dermatitis in all patients cleared with topical steroid. The relationship between positive patch testing and clinically relevant deep tissue reactions has not been delineated.

Lymphocyte transformation testing (LTT) or lymphocyte stimulation testing involves obtaining patient lymphocytes from a peripheral blood draw, and testing reactivity with a variety of antigens, including cobalt, nickel, and zirconium. Many argue that this test better replicates the sensitization that occurs in deep tissue after TJA, but its correlation to outcomes after arthroplasty has never been shown. Niki et al preformed lymphocyte stimulating testing on 92 patients (108 knees) undergoing primary TKA. 24 patients tested positive for metal hypersensitivity. Ultimately only five went on to develop dermatitis. Thus the clinical significance of positive results of lymphocyte stimulation testing is still unknown.

Additionally, serum metal levels are often elevated in patients with well-functioning TKA, and thus this test is not recommended for diagnosis of metal sensitivity. As a result, other causes such as infection, malalignment, aseptic loosening, referred pain, or systemic pain syndromes should all evaluated in persistently painful TKA.

At this time, metal sensitivity is not considered a significant cause of TKA failure. As the literature is inconclusive on identification and management of patients with metal hypersensitivity there is currently no indication for metal allergy screening prior to TKA. No study has found that patients with a previously known metal sensitivity have an increase rate of failure or revision TKA compared to those without. None of the major academic orthopedic societies recommend routine use of nickel free implants. There is currently no data showing correlation between nickel allergy and poor outcomes after total joint replacement with nickel containing implants. While non-nickel containing TKA implants have been developed, there is no evidence-based criteria for their use in specific patient populations. The goal of this study is to compare Knee Society Scores in patients with self-reported metal allergy who receive standard of care nickel containing implants vs oxidized zirconium nickel free implants for primary TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary TKA for the diagnosis of osteoarthritis or inflammatory arthritis with self-reported nickel allergy. Patients are routinely asked about nickel sensitivity as a part of the standard pre operative questionnaire already in place.

Exclusion Criteria:

* Patients less than 18 years of age
* Patients undergoing revision TKA
* Non english speaking patients
* Patient who have medical comorbidities that prevent elective TKA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | 3 weeks
  Change from pre operative to post operative Knee Society Scores at various time intervals. KSS is scored 0-100 with 100 being a perfectly functioning knee and is used as a gauge of success for a knee replacement.
Knee Society Score (KSS) | 6 weeks
  Change from pre operative to post operative Knee Society Scores at various time intervals. KSS is scored 0-100 with 100 being a perfectly functioning knee and is used as a gauge of success for a knee replacement.
Knee Society Score (KSS) | 1 year
  Change from pre operative to post operative Knee Society Scores at various time intervals. KSS is scored 0-100 with 100 being a perfectly functioning knee and is used as a gauge of success for a knee replacement.
Knee Society Score (KSS) | 2 years
  Change from pre operative to post operative Knee Society Scores at various time intervals. KSS is scored 0-100 with 100 being a perfectly functioning knee and is used as a gauge of success for a knee replacement.
Knee Society Score (KSS) | 5 years
  Change from pre operative to post operative Knee Society Scores at various time intervals. KSS is scored 0-100 with 100 being a perfectly functioning knee and is used as a gauge of success for a knee replacement.
Knee Society Score (KSS) | 10 years
  Change from pre operative to post operative Knee Society Scores at various time intervals. KSS is scored 0-100 with 100 being a perfectly functioning knee and is used as a gauge of success for a knee replacement.

SECONDARY OUTCOMES:
Complications | 90 days
  Any peri- or postoperative complications will be recorded including DVT/PE, return to the OR within 90 days, readmission within 90 days, superficial infection, deep infection, dermatitis, periprosthetic fracture, cerebrovascular accident/transient ischemic attack.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | 3 weeks
  Postoperative Knee Injury and Osteoarthritis Outcome Scores (KOOS JR) will also be recorded. This score is 0-100 with 100 being a perfectly functioning knee.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | 6 weeks
  Postoperative Knee Injury and Osteoarthritis Outcome Scores (KOOS JR) will also be recorded. This score is 0-100 with 100 being a perfectly functioning knee.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | 1 year
  Postoperative Knee Injury and Osteoarthritis Outcome Scores (KOOS JR) will also be recorded. This score is 0-100 with 100 being a perfectly functioning knee.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | 2 years
  Postoperative Knee Injury and Osteoarthritis Outcome Scores (KOOS JR) will also be recorded. This score is 0-100 with 100 being a perfectly functioning knee.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | 5 years
  Postoperative Knee Injury and Osteoarthritis Outcome Scores (KOOS JR) will also be recorded. This score is 0-100 with 100 being a perfectly functioning knee.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | 10 years
  Postoperative Knee Injury and Osteoarthritis Outcome Scores (KOOS JR) will also be recorded. This score is 0-100 with 100 being a perfectly functioning knee.
Radiographic assessment for proper component alignment and any signs of loosening | 3 weeks
  In addition, routine radiographs (AP and lateral knee radiographs) will be obtained at follow-up visits and assessed for component alignment and signs of loosening.
Radiographic assessment for proper component alignment and any signs of loosening | 6 weeks
  In addition, routine radiographs (AP and lateral knee radiographs) will be obtained at follow-up visits and assessed for component alignment and signs of loosening.
Radiographic assessment for proper component alignment and any signs of loosening | 1 year
  In addition, routine radiographs (AP and lateral knee radiographs) will be obtained at follow-up visits and assessed for component alignment and signs of loosening.
Radiographic assessment for proper component alignment and any signs of loosening | 2 years
  In addition, routine radiographs (AP and lateral knee radiographs) will be obtained at follow-up visits and assessed for component alignment and signs of loosening.
Radiographic assessment for proper component alignment and any signs of loosening | 5 years
  In addition, routine radiographs (AP and lateral knee radiographs) will be obtained at follow-up visits and assessed for component alignment and signs of loosening.
Radiographic assessment for proper component alignment and any signs of loosening | 10 years
  In addition, routine radiographs (AP and lateral knee radiographs) will be obtained at follow-up visits and assessed for component alignment and signs of loosening.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No